CLINICAL TRIAL: NCT04007198
Title: A Phase 1b Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of EQ001 in Subjects With Moderate-to-Severe Uncontrolled Asthma
Brief Title: A Study of Itolizumab (EQ001) to Evaluate the Safety, Tolerability, PK, PD, and Clinical Activity in Uncontrolled Asthma
Acronym: EQUIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Equillium (Industry)
Collaborators: Biocon Limited (Industry); Equillium AUS Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQ001-19-001
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: moderate-to-severe asthma
MeSH Terms: conditions — Asthma | interventions — itolizumab

STUDY DESIGN:
Intervention Model Description: up to 5 cohorts of 8 patients randomized 3:1 with ascending doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study site, participant and most vendors will be blinded. The site's pharmacist or designee will be unblinded to prepare the study drug. Relevant vendors including PK will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EQ001 (Experimental): EQ001 administered in a blinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 5 doses.
  Interventions: Drug: EQ001
- EQ001 Placebo (Placebo Comparator): Placebo administered in a blinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 5 doses.
  Interventions: Drug: EQ001 Placebo

INTERVENTIONS:
Drug: EQ001 — Itolizumab [Bmab 600]
  Other Names: Bmab600; Itolizumab
  Arms: EQ001
Drug: EQ001 Placebo — EQ001 Placebo
  Arms: EQ001 Placebo

SUMMARY:
This is a multi-center study to evaluate the safety, tolerability, PK, PD, and clinical activity of itolizumab (EQ001) in subjects with moderate-to-severe asthma.

DETAILED DESCRIPTION:
The study will enroll up to 40 subjects, with up to 5 dose escalating cohorts of 8 patients enrolled in a 3:1 ratio. Subjects will receive either itolizumab or placebo administered subcutaneously every two weeks (over 8 weeks) for a total of 5 doses with 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, age ≥ 18 and ≤ 75 years
2. Has a documented clinical diagnosis of moderate-to-severe uncontrolled asthma requiring moderate- or high-dose inhaled CS (ICS; ≥ 250 mcg of fluticasone propionate twice daily or equipotent ICS daily dosage to a maximum of 2000 mcg/day of fluticasone propionate or equivalent) and one or more additional controller medications (inhaled LABA or anticholinergic or LTA) for ≥ 3 months, with a stable dose ≥1 month prior to the initial Screening Visit
3. Has a prebronchodilator forced expiratory volume in 1 second (FEV1) ≥ 40% and ≤ 90% of predicted value during the Screening Period, despite use of a moderate- or high-dose ICS and one or more additional controller medications (inhaled LABA or anticholinergic or LTA)
4. Has a history of clinically diagnosed asthma, which could include a history of FEV1 reversibility and/or positive bronchial challenge test
5. Has a history of ≥ 1 clinically significant asthma exacerbation prior to the initial Screening Visit, despite use of a moderate- or high dose ICS and one or more additional controller medications at the time the exacerbation(s) occurred

Exclusion Criteria:

1. Is a current or former smoker with a smoking history of ≥10 pack-years (number of pack-years = number of cigarettes per day/20 × number of years smoked; a former smoker is defined as a subject who stopped smoking ≥ 6 months prior to the Screening Visit)
2. Has a body mass index > 36 kg/m2
3. Has a documented history or radiological evidence of a clinically important lung condition other than asthma (eg, α1 antitrypsin deficiency, bronchiectasis, cystic fibrosis, primary ciliary dyskinesia, pulmonary fibrosis, allergic bronchopulmonary mycosis, or lung cancer)
4. Has a respiratory tract infection (RTI) within 4 weeks before the initial Screening Visit, or during the Screening Period (these subjects may be re-screened following complete resolution of their RTI)
5. Has an asthma exacerbation within 4 weeks before the initial Screening Visit, or during the Screening Period (these subjects may be re-screened following complete resolution of their exacerbation)
6. Has a diagnosis of currently active malignancy; subjects with a medical history of basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the uterine cervix are eligible; subjects with a medical history of other malignancies are eligible if the subject is in remission and curative therapy was completed ≥ 2 years prior to the initial Screening Visit
7. Has a history or presence of clinically concerning cardiac arrythmias, atrial fibrillation, New York Heart Association Class III or IV heart failure, or prolonged QT or corrected QT interval > 500 milliseconds (ms) at the Screening Visit
8. Has any disorder (including, but not limited to, cardiovascular [CV], gastrointestinal [GI], hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment) that is not stable in the opinion of the investigator and/or could:

   1. Affect the subject's safety
   2. Influence the findings of the study or data interpretation
   3. Impede the subject's ability to complete the study
9. Has undergone bronchial thermoplasty
10. Has a history of substance abuse (including alcohol) that may, in the investigator's judgment, increase the risk to the subject of participation in the study
11. Has used monoclonal antibody (mAb) therapy for the management of asthma or any other condition within 3 months prior to the initial Screening Visit (these subjects may be re-screened following the 3 month period)
12. Has required an oral corticosteroid burst within 1 month prior to the initial Screening Visit or during the Screening Period (these subjects may be re-screened following the 1 month period); maintenance oral corticosteroids ≤ 10 mg/d prednisone or equivalent is permitted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo A Douglass, MD, Principal Investigator — Melbourne Health
Locations (13):
- Australia (9):
  - Flinders Medical Centre, Adelaide
  - Box Hill Hospital, Box Hill
  - Monash Medical Centre, Clayton
  - Paratus Clinical Research Central Coast, Kanwal
  - Respiratory Clinical Trials, Kent Town
  - TrialsWest, Murdoch
  - Melbourne Health, Parkville
  - Paratus Clinical Research Western Sydney, Sydney
  - The Queen Elizabeth Hospital, Woodville
- New Zealand (4):
  - Respiratory Research, Greenland Clinical Centre, Auckland
  - Dunedin Hospital, Dunedin
  - The New Zealand Respiratory & Sleep Institute, Greenlane
  - Medical Research Institute of New Zealand, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: company website — https://equilliumbio.com/
- See also: Australia New Zealand Clinical Trials Registry — http://www.anzctr.org.au/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts for dose 2.4mg/kg and 3.2mg/kg were not conducted. Data for placebo subjects in cohort for 0.8mg/kg and 1.6mg/kg were pooled in analysis.
Groups:
- EQ001 0.8mg/kg: EQ001 administered in a blinded fashion by subcutaneous injection every two weeks for a total of 5 doses at 0.8mg/kg EQ001: Itolizumab [Bmab 600]
- EQ001 Placebo: EQ001 Placebo administered in a blinded fashion by subcutaneous injection every two weeks for a total of 5 doses.
  EQ001 Placebo: EQ001 Placebo
- EQ001 1.6mg/kg: EQ001 administered in a blinded fashion by subcutaneous injection every two weeks for a total of 5 doses at 1.6mg/kg EQ001: Itolizumab [Bmab 600]
Period: Overall Study
Arm/Group | EQ001 0.8mg/kg | EQ001 Placebo | EQ001 1.6mg/kg
Started | 7 | 4 | 7
Completed | 6 | 4 | 6
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- EQ001 0.8mg/kg: EQ001 administered in a blinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 5 doses at 0.8mg/kg.
  EQ001: Itolizumab [Bmab 600]
- EQ001 1.6mg/kg: EQ001 administered in a blinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 5 doses at 1.6mg/kg.
  EQ001: Itolizumab [Bmab 600]
- Total: Total of all reporting groups
Arm/Group | EQ001 0.8mg/kg | EQ001 Placebo | EQ001 1.6mg/kg | Total
Number analyzed (Participants) | 7 | 4 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (15.59) | 56.0 (6.73) | 50.1 (18.53) | 52.2 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 4 | 2 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 4 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 1 | 2
  Australia | 6 | 4 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: Study Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | EQ001 0.8mg/kg | EQ001 Placebo | EQ001 1.6mg/kg
Number analyzed (Participants) | 7 | 4 | 7
Participants | 6 | 1 | 7

2. Secondary Outcome: Time to Maximum EQ001serum Concentration, Tmax
Description: Time to maximum EQ001 serum concentration, Tmax
Time Frame: Study Day 85
Reporting Status: Not Posted

3. Secondary Outcome: Maximum EQ001 Serum Drug Concentration, Cmax
Description: Maximum EQ001 serum drug concentration, Cmax
Time Frame: Study Day 85
Reporting Status: Not Posted

4. Secondary Outcome: Minimum EQ001 Serum Drug Concentration, Cmin
Description: Minimum EQ001 serum drug concentration prior to next dose, Cmin
Time Frame: Study Day 85
Reporting Status: Not Posted

5. Secondary Outcome: Total EQ001 Exposure Across Time, AUC (From Zero to Infinity)
Description: Total EQ001 exposure across time, AUC (from zero to infinity)
Time Frame: Study Day 85
Reporting Status: Not Posted

6. Secondary Outcome: Volume of Distribution of EQ001, Vd
Description: Volume of distribution of EQ001, Vd
Time Frame: Study Day 85
Reporting Status: Not Posted

7. Secondary Outcome: Clearance, Cl
Description: Clearance, Cl
Time Frame: Study Day 85
Reporting Status: Not Posted

8. Secondary Outcome: Inflammatory Markers
Description: Including but not limited to: IL-1β, IL-2, IL-6, IL-17, IL-21, IL-22, IL-23, IFN-γ, and TGF-β, C-reactive protein
Time Frame: Study Day 85
Reporting Status: Not Posted

9. Secondary Outcome: CD6 Receptor Expression
Description: the % levels of free versus EQ001-bound CD6 receptor on T cells
Time Frame: Study Day 85
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time Frame: Study Day 85
Groups:
- EQ001 0.8mg/kg: EQ001 administered in a blinded fashion by subcutaneous injection every two weeks for a total of 5 doses at 0.8mg/kg.
  EQ001: Itolizumab [Bmab 600]
- EQ001 1.6mg/kg: EQ001 administered in a blinded fashion by subcutaneous injection every two weeks for a total of 5 doses at 1.6mg/kg.
  EQ001: Itolizumab [Bmab 600]
Arm/Group | EQ001 0.8mg/kg | EQ001 1.6mg/kg | EQ001 Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 0/4
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 0.8mg/kg (N=7) | EQ001 1.6mg/kg (N=7) | EQ001 Placebo (N=4)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 0.8mg/kg (N=7) | EQ001 1.6mg/kg (N=7) | EQ001 Placebo (N=4)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 0 (0)
Injection site reaction (General disorders) | 4 (4) | 2 (2) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT04007198/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT04007198/SAP_001.pdf